CLINICAL TRIAL: NCT06984887
Title: An Evaluation of New TB Diagnostic Tests (NATs) for Active Case Finding for TB in Pakistan
Brief Title: Evaluation of New TB Diagnostic Tests (NATs) in Pakistan
Acronym: TB
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Corps Pakistan (Other)
Collaborators: Centre for Global Public Health Pakistan (Other); Royal Tropical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INV-045723
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis Diagnosis
Keywords: New TB diagnostics; New NATs for TB; Cost efficient TB diagnostic tools
MeSH Terms: interventions — Diagnostic Techniques and Procedures

STUDY DESIGN:
Intervention Model Description: A diagnostic non-inferiority trial design will be followed to demonstrate that the new diagnostic tests (NAT) is equal to/not lesser than the existing standard test (Xpert MTB/Rif Assay).
  The aim of this trial is not to prove that the new test is better, but to show that the performance of the new tests is comparable to the current test which is used in ACF settings in Pakistan. The two new, the reference diagnostic test (Xpert Ultra) and the gold standard test (MTB culture) will be done in parallel to allow for a direct comparison of the two new tests and the reference test, performed on the same set of samples from each participant. This diagnostic evaluation study is cross-sectional in nature as it will typically involve assessing a diagnostic test's performance (such as sensitivity, specificity, etc.) at a single point in time. The key outcomes will be assessed using culture-confirmed TB and culture negative TB as a reference standard.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic Trial (Experimental)
  Interventions: Diagnostic Test: Diagnostic procedures

INTERVENTIONS:
Diagnostic Test: Diagnostic procedures — This study will be evaluated by conducting a non-inferiority diagnostic trial within routine ACF settings by comparing the New Diagnostic tests (NAT) to the reference standard test (Xpert MTB/Rif Assay) to determine how well it can detect and diagnose TB. All samples will be tested for MTB using cultures.

SUMMARY:
This study aims to test new diagnostic methods for tuberculosis (TB) testing as compared to the existing Xpert MTB/Rif Ultra testing approach. The research questions that will be addressed by this study include:

* What are the sensitivity and specificity of the new diagnostic tests Pluslife MTBC and Ustar PortNAT for tuberculosis and how do these compare to Xpert Ultra?
* How does the new diagnostic method compare to Xpert Ultra in terms of implementation feasibility, cost and turnaround time?
* What are the logistical and technical advantages and challenges associated with implementing the new diagnostic method compared to Xpert Ultra?
* What are the perceptions of healthcare providers as well as sample provider regarding the usability, feasibility and convenience of use of the new sample collection method compared to existing methods?

DETAILED DESCRIPTION:
Research Objective 1:

The study aims to assess the diagnostic accuracy-specifically the sensitivity and specificity-of two new NAT-based tuberculosis (TB) tests, Pluslife and Ustar. These tests will be compared against the existing reference standard, the Xpert MTB/Rif Ultra, with culture testing used as the gold standard. This evaluation will take place in the context of Active Case Finding (ACF) in Pakistan. The research will follow a non-inferiority diagnostic trial design. The procedure involves testing all samples with cultures and comparing the results from the new NAT tests against the reference to determine their effectiveness in detecting and diagnosing TB.

Expected Outcomes:

Sensitivity of the new NAT tests Specificity of the new NAT tests False positive rate False negative rate

Research Objective 2:

This objective focuses on evaluating the operational feasibility, cost-effectiveness, and turnaround time of the new NAT diagnostics compared to the Xpert Ultra platform. The strategy will involve both quantitative and qualitative research methods. Quantitative data will be collected and analyzed regarding the cost per test and the time taken from sample receipt to result reporting. In addition, a qualitative study will be conducted using semi-structured in-depth interviews with presumptive TB patients and healthcare providers involved in sample collection at ACF camp settings. These interviews will explore experiences, challenges, and preferences related to the use of sputum samples versus tongue swabs.

Expected Outcomes:

Cost per test performed Average turnaround time for each NAT platform Preferences of sample providers regarding collection methods Preferences of healthcare providers regarding sample collection methods Specific challenges associated with each collection method Barriers to compliance with sample collection Overall feasibility and ease of use of the diagnostic approaches

Research Objective 3:

The third objective seeks to assess the acceptability and usability of tongue swab-based sample collection compared to traditional sputum sample methods. This will be explored through a qualitative inquiry, gathering in-depth insights from both sample providers and healthcare workers to understand their perspectives, experiences, and any usability issues associated with each method.

Expected Outcomes:

Insights into user and provider acceptance of tongue swab versus sputum collection Identification of usability challenges and practical considerations in sample collection methods

ELIGIBILITY:
Inclusion Criteria:

* People who are screened for TB on X-ray with CAD and their CAD scores are available
* Age range appropriate for the test (e.g., adult patients 12 yrs old and above)
* Any gender
* Consent to participate in the study and provide samples (e.g., tongue swab, sputum).

Exclusion Criteria:

* Pregnant women (depending on the diagnostic method or potential risks involved).
* Known cases of Pulmonary TB
* People who are unable to produce sputum
* Extra Pulmonary TB cases
* People who are not screened for TB on X-ray and/or their CAD scores are not available

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6100 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with positive and negative Mycobacterium Tuberculosis | From enrolment to the end of results confirmation at 8 weeks
  The results of each of the test performed (negative and positive TB) using Pluslife MTBC test result, Ustar's PortNAT test result, Xpert MTB/Rif test result and results of the MTB culture.

CONTACTS AND LOCATIONS:
Locations (1):
- National Reference Laboratory, Islamabad, Federal Capital, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided